CLINICAL TRIAL: NCT00048620
Title: Double-Blind,2 Dose Group Study of Recombinant Human N-Acetylgalactosamine 4-Sulfatase in Patients With MPS VI
Brief Title: Study of Recombinant Human N-Acetylgalactosamine 4-Sulfatase in Patients With MPS VI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASB-00-01
Record Dates: First submitted 2002-11-04; First posted 2002-11-06 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2006-11

CONDITIONS: Mucopolysaccharidosis VI
MeSH Terms: conditions — Mucopolysaccharidosis VI | interventions — N-Acetylgalactosamine-4-Sulfatase

INTERVENTIONS:
Drug: N-acetylgalactosamine 4-sulfatase

SUMMARY:
The purpose of the study is to evaluate the safety, efficacy and pharmacokinetics of two dose levels of weekly intravenous infusions of recombinant human N-acetylgalactosamine 4-sulfatase (rhASB) for a minimum of 24 weeks in patients diagnosed with MPS VI.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Patient must be five years of age or older
* Patient must have documented diagnosis of MPS VI, confirmed at screening by measurable clinical signs and symptoms of MPS VI
* Leukocyte ASB enzyme activity level less than 20% of the normal range
* Clinical evidence of significant MPS VI disease that provides adequate opportunity to achieve quantitative, short-term therapeutic benefit in three or more of the following parameters: endurance (as measured by a six-minute walk test), forced vital capacity (as measured by spirometry), joint range of motion, urinary glycosaminoglycans, and hepatomegaly.
* Ability to perform all protocol tests
* Ability to stand independently for six minutes
* Sexually active subjects must agree to use an adequate form of contraception

Exclusion Criteria:

* History of bone marrow transplantation
* Pregnant or lactating patient
* Use of an investigational drug or device within 30 days prior to study participation.
* A medical condition, serious intercurrent illness, or other extenuating circumstances that may significantly decrease study compliance including prescribed follow-up
* Known hypersensitivity to rhASB or to components of the study drug
* History of cancer (except low grade and fully resolved skin malignancy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Study Completion 2005-11

PRIMARY OUTCOMES:
Lysosomal storage disease

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Swiedler, MD, Ph.D., Study Director — BioMarin Pharmaceutical
Locations (1):
- BioMarin Pharmaceutical Inc., Novato, California, United States

REFERENCES:
- See also: Related Info — http://www.bmrn.com